CLINICAL TRIAL: NCT06045663
Title: Cervical Laminectomy With or Without Lateral Mass Fixation in Cervical Spondylotic Myelopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Moustafa ElBadry Alrabyi Ahmed, Resident of neurosurgery department, Sohag University Hospitals, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-09-02MS
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Cervical Myelopathy (DCM)
MeSH Terms: interventions — Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- laminectomy group (Active Comparator): patient will divided into two group the first group will undergo cervical laminectomy while the second group will undergo cervical laminectomy with lateral mass fixation .all surgical related events and comorbidities will be recorded.
  the patient will examine after 3 months of operation and patient's myelopathy grade and functional status was evaluated after 6 months using modified Japanese orthopedic association (mJAO) score. Radiological Follow-up by using plain X-rays, 6 months follow up assessment of cervical spine sagittal alignment using (C2-C7) Cobb's angle and MRI scan if needed follow up will be at our department follow up clinic .
  Interventions: Procedure: laminectomy without lateral mass fixation
- laminectomy with lateral mass fixation (Active Comparator): patient will divided into two group the first group will undergo cervical laminectomy while the second group will undergo cervical laminectomy with lateral mass fixation .all surgical related events and comorbidities will be recorded.
  the patient will examine after 3 months of operation and patient's myelopathy grade and functional status was evaluated after 6 months using modified Japanese orthopedic association (mJAO) score. Radiological Follow-up by using plain X-rays, 6 months follow up assessment of cervical spine sagittal alignment using (C2-C7) Cobb's angle and MRI scan if needed follow up will be at our department follow up clinic .
  Interventions: Procedure: laminectomy with lateral mass fixation

INTERVENTIONS:
Procedure: laminectomy without lateral mass fixation — patient will divided into two group the first group will undergo cervical laminectomy without lateral mass fixation while the second group will undergo cervical laminectomy with lateral mass fixation while the second group will undergo cervical laminectomy with lateral mass fixation
  Arms: laminectomy group
Procedure: laminectomy with lateral mass fixation — patient will divided into two group the first group will undergo cervical laminectomy without lateral mass fixation while the second group will undergo cervical laminectomy with lateral mass fixation while the second group will undergo cervical laminectomy with lateral mass fixation
  Arms: laminectomy with lateral mass fixation

SUMMARY:
The cervical spine consists of seven cervical vertebrae joined by intervertebral disks and a complex network of ligaments. The cervical spine has a normal lordotic curve, and it is much more mobile than the thoracic or lumbar regions of the spine, which makes it more liable to both degenerative and traumatic disorders .

Degenerative cervical myelopathy (DCM) is the most common form of spinal cord dysfunction in adults. The incidence and prevalence of myelopathy due to degeneration of the spine are estimated at a minimum of 41 and 605 per million in North America and Incidence of cervical spondylotic myelopathy-related hospitalizations has been estimated at 4.04/100,000 person-years.

Degenerative cervical myelopathy (DCM), earlier referred to as cervical spondylotic myelopathy, Patients report neurological symptoms such as pain and numbness in limbs, poor coordination, imbalance, and bladder dysfunction.

Surgical management for patients with multilevel cervical myelopathy aims to decompress the spinal cord and restore the normal sagittal alignment using either an anterior approach or a posterior approach. Multilevel anterior surgery is associated with complications such as increased surgical trauma and increased incidence of pseudarthrosis, graft dislodgement, and implant failure as the number of level increases.The posterior approach is optimal for multilevel stenosis using consecutive laminectomies However, although the effectiveness of cervical laminectomy was documented repeatedly, there were still concerns over postoperative kyphotic deformity, cervical instability, and late deterioration Cervical laminectomy and fusion may be performed to avoid the potential complications of instability and kyphosis associated with cervical laminectomy alone. For the latter, dissection and removal of the posterior elements disrupts the normal biomechanics of the cervical spine, leading to post laminectomy deformity and instability Our study aim to evaluate the multilevel cervical laminectomy alone, and multilevel cervical laminectomy with lateral mass fixation in patients with cervical spondylotic myelopathy regarding the Clinical and radiological outcome for short term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms of spondylotic myelopathy at two or more level cervical canal stenosis after full filling clinical and radiological criteria

Exclusion Criteria:

* History of previous cervical intervention like (anterior cervical approach and laminoplasty ).
* History of cervical trauma.
* History of other neurological disorders such as( Multiple sclerosis , stroke,AML,….ETC).
* patient with insuffient data.
* Uncontrolled DM, hypertension and thyroid disorders.
* Osterpenic or osteoporotic patients

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
assessment of cervical spine sagittal alignment | 6 months
  assessment of cervical spine sagittal alignment using (C2-C7) Cobb's angle

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohamed E, Ihab Z, Moaz A, Ayman N, Haitham AE. Lateral mass fixation in subaxial cervical spine: anatomic review. Global Spine J. 2012 Mar;2(1):39-46. doi: 10.1055/s-0032-1307261. PMID 24353945
- [Background] Singrakhia MD, Malewar NR, Singrakhia SM, Deshmukh SS. Cervical Laminectomy with Lateral Mass Screw Fixation in Cervical Spondylotic Myelopathy: Neurological and Sagittal Alignment Outcome: Do We Need Lateral Mass Screws at each Segment? Indian J Orthop. 2017 Nov-Dec;51(6):658-665. doi: 10.4103/ortho.IJOrtho_266_16. PMID 29200481